CLINICAL TRIAL: NCT05491356
Title: The Utility of Intra-Catheter Fibrinolytics in Draining Chronic Subdural Hematomas: A Randomized Controlled Trial Pilot Study
Brief Title: Use of Tissue Plasminogen Activator in the Clearance of Chronic Subdural Hematomas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14724
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2024-03

CONDITIONS: Hematoma, Subdural; Fibrinolytic; Hemorrhage
MeSH Terms: conditions — Hematoma, Subdural; Hemorrhage | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - tPA administered (Experimental): This group will receive 2mL of intra-catheter tPA during twist drill craniostomy procedure
  Interventions: Drug: Tissue Plasminogen Activator
- Placebo Control (Placebo Comparator): This group will receive 2mL of intra-catheter saline solution during twist drill craniostomy procedure
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tissue Plasminogen Activator — Dosage of 1mg/mL mixed in 0.9% saline solution, intra-catheter administration, sterile
  Arms: Intervention - tPA administered
Drug: Placebo — 0.9% saline solution, intra-catheter administration, sterile
  Arms: Placebo Control

SUMMARY:
To determine the utility of tissue plasminogen activator (tPA) in the clearance of chronic subdural hematomas (CSDH). Intra-catheter tPA will be administered during surgical procedure and allowed to break down blood clot to assist with removal/drainage during twist drill craniostomy procedure.

DETAILED DESCRIPTION:
A chronic subdural hematoma (CSDH) is a collection of blood overlying the brain that can be seen, usually in the elderly with even minimal head trauma. These are usually treated by removing the collection of blood. This can be done through a small drill hole in the skull or by larger holes (one or two) the size of a nickel. Sometimes a larger piece of skull is removed to be able to remove the CSDH. The standard practice at our center is to do these procedures under local anesthesia with a twist drill craniostomy (small drill hole through the skull). In some cases, all the CSDH can not be removed the first time, requiring a second procedure or a larger procedure. This study plans to use a type of medication that breaks down the solid blood clot, enabling more of it to drain. This medication (tpa) is already used in other surgeries and is safe to use in humans. Our preliminary experience and that of others suggests very low risk at the dosages being used. We hope that using this new drug will decrease the chance of the CSDH collecting again and reduce the overall length of your stay in the hospital and reduce the need for further surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (18 yrs or older)
2. Admitted to neurosurgery wing at the hospital
3. Symptomatic patients requiring surgical drainage by twist drill craniostomy

Exclusion Criteria:

1. Patients at increased risk of bleeding such as patients taking anticoagulation medication that required reversal at time of intervention، or those with coagulopathic disorder.
2. Patients on antiplatelets or anticoagulation medications (DOACs or warfarin) with appropriate holding period prior to drainage, those who are eventually minimized to a regular bleeding risk compared to the normal population, will be included in the study.
3. Patients with subdural empyema.
4. Redo twist drill craniostomy for residual cSDH within the same admission.
5. Drain accidentally removed during nursing care or patient transport before 24 hr interval scan.
6. Patients who are not expected to live more than three months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Study Feasibility | 8 months
  Patient recruitment rate, eligibility of patients, protocol adherence, unexpected events

SECONDARY OUTCOMES:
Reoperation rate | 8 months
  Reoperation rate in the first 6 weeks post drainage
Volume of chronic subdural hematoma | 8 months
  Volume, as measured in 3 intervals: pre-procedure, post-procedure at 24hrs and 6 weeks
Rate of adverse events | 8 months
  Rate of adverse events in the first 6 weeks post procedure, including CNS infection, seizure, post-op hemorrhage
Length of hospital stay | 8 months
  length of hospital stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Kesava Reddy, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
Patient data will be de-identified and the data will be analyzed as a whole before becoming available to other researchers.
  De-identified IPD may be shared with other researchers if necessary based on occurrence of adverse events occurrence, circumstantial findings, etc.

REFERENCES:
- [Background] Neils DM, Singanallur PS, Wang H, Tracy P, Klopfenstein J, Dinh D, Elwood PW, Fassett D, McCall T, Lin J, Tsung A. Recurrence-free chronic subdural hematomas: a retrospective analysis of the instillation of tissue plasminogen activator in addition to twist drill or burr hole drainage in the treatment of chronic subdural hematomas. World Neurosurg. 2012 Jul;78(1-2):145-9. doi: 10.1016/j.wneu.2011.08.032. Epub 2011 Nov 7. PMID 22120294
- [Background] Brazdzionis J, Patchana T, Wiginton JG 4th, Wacker MR, Menoni R, Miulli DE. Intracatheter Tissue Plasminogen Activator for Chronic Subdural Hematomas after Failed Bedside Twist Drill Craniostomy: A Retrospective Review. Cureus. 2019 Dec 26;11(12):e6472. doi: 10.7759/cureus.6472. PMID 32025399
- [Background] O YM, Tsang SL, Leung GK. Fibrinolytic-Facilitated Chronic Subdural Hematoma Drainage-A Systematic Review. World Neurosurg. 2021 Jun;150:e408-e419. doi: 10.1016/j.wneu.2021.03.029. Epub 2021 Mar 17. PMID 33722722